CLINICAL TRIAL: NCT01919840
Title: Indicación de transfusión de Hemoderivados en el Postoperatorio de cirugía Cardiaca Tras la implantación de un Sistema de monitorización de la coagulación a la Cabecera Del Paciente: Tromboelastometría Versus Protocolo Habitual de transfusión
Brief Title: Blood Products Transfusion in Cardiac Surgery After the Implementation of a Coagulation Monitoring System at Patient Bedside: Thromboelastometry Versus Standard Transfusion Protocol
Acronym: ROTEM-2010
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment after the expected time to finish the study
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIBSP-ROT-2010-15
Record Dates: First submitted 2013-04-12; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Hemostatic Disorders
Keywords: hemostatic disorders; ardiac surgery; cardiopulmonary bypass
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group C (Active Comparator): • conventional protocol, volume replacement with massive bleeding.
  Interventions: Other: Group C
- Group ROTEM (Experimental): • Protocol according to the different tests to be performed with thromboelastography
  Interventions: Procedure: Group ROTEM

INTERVENTIONS:
Procedure: Group ROTEM — 10 min after administration of protamine, if there is a large diffuse microvascular bleeding or bleed excessively at the exit of surgery then will check an Intem, a Heptem a Extem and Fibtem.
  If any of the determinations altered and the patient leaves still bleeding apply the proposed treatment algorithm for Rotem. 10 minutes after each treatment will take the test again indicated that treatment, to ensure that the defect has been corrected.
  Arms: Group ROTEM
Other: Group C — 10 min. after protamine administration, if there is a significant diffuse microvascular bleeding or when the patient departure from surgery if bleeds excessively will be a TCA and routed the following analytical results: prothrombin time, activated partial thromboplastin time, platelet count and fibrinogen.
  If any of the determinations altered and the patient still bleeding, apply the standard protocol of the unit. 10 minutes after each treatment was performed new laboratory tests to analyze the result.
  Arms: Group C

SUMMARY:
Main objective:

Determine whether by introducing thromboelastograph, the investigators reduced the number of packed red cells received by each patient (median) compared to the usual protocol, in which the indication for transfusion is based on laboratory tests: Prothrombin time, time activated partial thromboplastin time, thrombin, reptilase, fibrinogen and platelet contage.

Design:

Prospective randomized controlled trial and single blinded.

Disease or disorder under study:

Study of coagulopathy in patients undergoing cardiac surgery with cardiopulmonary bypass (CPB).

Primary endpoint:

median transfusion of packed red blood cells per patient. Study population Male and female patients over 18 years undergoing cardiac surgery with cardiopulmonary bypass to bleed excessively.

Duration of treatment:

The coagulation monitoring methods tested are made from protamine administration to CEC output if a) the patient bleeds diffusely, or b) from arrival in the unit if not satisfied critics a) bleed excessively drains and until the patient stops bleeding (debit drains <a 150ml / h).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* over 18 years
* undergoing cardiac surgery
* with cardiopulmonary bypass
* bleed excessively

As it is not possible to predict in advance who will bleed, informed consent will be required for all patients over 18 who are to undergo cardiac surgery with CPB.

Will be randomized to either group

1. Those patients with diffuse bleeding after protamine administration. and / or
2. They bleed excessively after surgery. Are excessive bleeding criteria: the debit ≥ 300ml drains in the first hour; ≥ 250ml in the second hour or ≥ 150ml at any later time. Consider that the patient is bleeding excessively when the drains debit is <150ml.

Exclusion Criteria:

* Patients <18 years
* Extracorporeal circulation surgery
* Surgery with Mini extracorporeal circulation (MECC)
* Refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
median transfusion of packed red cells per patient | 24 hours

SECONDARY OUTCOMES:
rate transfusion of platelets pool and plasma pool | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Paniagua, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau